CLINICAL TRIAL: NCT06971991
Title: qDSA Blood Flow Measurement in Patients Undergoing Transarterial Embolization (TAE) of the Liver
Brief Title: qDSA Blood Flow Measurement in Patients Undergoing TAE of the Liver
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2024-1159; A539300 (Other: UW Madison); Protocol Version: 4/18/24 (Other: UW Madison)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Transarterial Embolism; Transarterial Chemoembolization
Keywords: Quantitative digital subtraction angiography (qDSA)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Participants Undergoing TAE of the Liver (Experimental)
  Interventions: Device: qDSA Blood Flow Measurement

INTERVENTIONS:
Device: qDSA Blood Flow Measurement — The research intervention is limited to several additional qDSA image acquisitions, which include administration of additional iodinated contrast medium.

SUMMARY:
The purpose of this research is to evaluate a new technique, quantitative digital subtraction angiography (qDSA), to measure blood flow during liver embolization procedures. Liver transarterial embolization is a way of treating liver tumors by blocking blood flow to it. The qDSA technique could help doctors ensure the blood flow to the tumor is decreased by the right amount by calculating blood flow before, during, and after the procedure. Up to 20 participants will be enrolled for 1 study visit and data collection for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary, written informed consent to participate in this study and willing to comply with study-related evaluation and procedure schedule

Exclusion Criteria:

* Pregnancy or breastfeeding
* Patients with an acute kidney injury or stage IV or V chronic kidney disease (Cr greater than 2.4 or estimated glomerular filtration rate (eGFR) less than 30), unless anuric and on dialysis without expected return of renal function.
* Patients with an iodinated contrast allergy who cannot be adequately premedicated to receive contrast as part of the embolization procedure.
* Patients with a physical or psychological condition that would impair study participation.
* The patient is judged unsuitable for study participation by the Investigator for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients in which qDSA measurements demonstrate successive reductions in hepatic arterial velocity at the pre-, mid-, and post-embolization time points | data collected pre-embolization, mid-embolization, and post-embolization (up to 1 hour), data processed retrospectively for this measure when data collection is complete (up to 6 months)

SECONDARY OUTCOMES:
Assessment of flow reductions using qDSA compared with conventional DSA (current clinical standard): Percent Flow reduction from baseline | data collected pre-embolization, mid-embolization, and post-embolization (up to 1 hour), data processed retrospectively for this measure when data collection is complete (up to 6 months)
  This will be done through a reader study where interventional radiologists will review conventional pre-, mid-, and post-embolization DSA sequences and asked to quantify the percent flow reduction relative to baseline.
Assessment of flow reductions using qDSA compared with conventional DSA (current clinical standard): Number of procedures retrospectively judged to end early | data collected pre-embolization, mid-embolization, and post-embolization (up to 1 hour), data processed retrospectively for this measure when data collection is complete (up to 6 months)
  This will be done through a reader study where interventional radiologists will review conventional pre-, mid-, and post-embolization DSA sequences and asked to judge whether the embolization procedure should proceed or end.
Velocity measurements made on qDSA vs transabdominal Doppler US | measured during transarterial embolism (up to 1 hour), qDSA data processed retrospectively when data collection is complete (up to 6 months)
  qDSA results (relative velocity drop as well as absolute velocities when possible) will be compared to transabdominal ultrasound measurements acquired during the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Laeseke, MD, PhD, Principal Investigator — UW School of Medicine and Public Health
Locations (1):
- UW Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
The study team will seek and IRB determination prior to any secondary uses of data in the future for research related to qDSA. A change of protocol will be submitted to the IRB to report any sharing of data to institutions other than the sponsor.